CLINICAL TRIAL: NCT07107945
Title: A Randomised, Double-blind, Placebo-controlled Trial With an Open-label Extension to Assess the Pharmacokinetics, Safety, and Efficacy of Empagliflozin Tablets in Paediatric Patients With Chronic Kidney Disease (EMPA-KIDNEY® Kids)
Brief Title: A Study to Find Out How EMPAgliflozin is Tolerated and if it Helps Children and Adolescents With Chronic KIDNEY Disease (EMPA-KIDNEY® Kids)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1245-0256; 2024-512577-27-00 (Registry Identifier: CTIS); U1111-1312-1389 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-08-05; First posted 2025-08-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin treatment arm (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Other Names: Jardiance
  Arms: Empagliflozin treatment arm
Drug: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
This study is open to children aged 2 to 17 with chronic kidney disease (CKD). The purpose of this study is to find out if a medicine called empagliflozin helps children and adolescents with CKD. Other goals of the study are to find out how empagliflozin is tolerated and handled by the body in children and adolescents with CKD.

Participants are put into 2 groups randomly, which means by chance. One group takes empagliflozin and the other group takes placebo. Placebo looks like empagliflozin but does not contain any medicine. Participants are twice as likely to be in the empagliflozin group. Participants take empagliflozin or placebo as tablets once a day for 6 months. After 6 months, participants in both groups take empagliflozin as tablets once a day for 1 year.

Participants are in the study for a little over a year and a half. During this time, they visit the study site about 15 times and get at least 5 phone or video calls from the site staff. At the visits, the doctors take blood and urine samples from the participants. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent provided by the patient's parent(s) (or legal guardian) and patient's assent in accordance with international council for harmonisation good clinical practice (ICH-GCP) and local legislation prior to admission to the trial (informed assent will be sought according to the patient's age, level of maturity, competence, and capacity).
* Age 2 to 17 years at screening Visit 1.
* Chronic kidney disease (CKD) of any underlying aetiology defined by (as measured by central laboratory at screening Visit 1): estimated glomerular filtration rate (eGFR) (U25Crea) ≥20 to <90 mL/min/1.73 m2 with a urine-albumine-creatinine (UACR) ≥300 mg/g
* Participants must be on a stable dose of maximally tolerated standard of care (SoC) therapy for 30 days before screening visit 1 with no plans to change the dose throughout the duration of the placebo-controlled duration of the trial. SoC is anticipated to include a single Renin-angiotensin-aldosterone system (RAAS) inhibitor, such as angiotensin receptor blockers (ARB) or angiotensin converting enzyme inhibitors (ACEi) as appropriate and tolerated. Additional use of a mineralocorticoid receptor antagonist (MRA, including finerenone if available) is permitted if needed and the dose is stable for 30 days before screening Visit 1 and no planned dose changes for the placebo-controlled portion of the trial.
* Participants receiving daily immunosuppressive therapy for an underlying immunological cause of CKD must be on a stable dose for the duration specified for each drug prior to screening and must remain on a stable regimen throughout the placebo-controlled portion of the trial.
* Further inclusion criteria apply.

Exclusion Criteria:

* Confirmed type 1 or type 2 diabetes mellitus.
* History of ketoacidosis within 8 weeks prior to Visit 1 and up to randomisation.
* Chronic dialysis or functioning kidney transplant or scheduled for transplantation throughout the duration of the trial.
* Diagnosis of uncontrolled metabolic bone disease (at the Investigator's discretion).
* Body mass index (BMI) ≤10th percentile for children ≥4 years of age and ≤25th percentile for children <4 years of age according to Centers for Disease Control and Prevention (CDC) growth chart at screening Visit 1.
* Gastrointestinal disorders that might interfere with trial drug absorption according to investigator assessment.
* Presence of acute or active urinary tract infection (UTI) with signs or symptoms of an active UTI or therapeutic treatment for an active UTI within 14 days before screening Visit 1.
* Severe, uncontrolled hypertension (based on investigator's judgement).
* Further exclusion criteria apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-06-26 (Estimated); Study Completion 2029-06-25 (Estimated)

PRIMARY OUTCOMES:
Change from Day 1 to the Week 24 visit in urine albumin-creatinine (UACR) [mg/g] | Up to week 24
Change from Day 1 to the Week 24 visit in urine glucose [mmol/L] | Up to week 24

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) (U25Crea) over time during treatment with empagliflozin | Up to week 73
  U25Crea = estimates the glomerular filtration rate based on creatinine in patients aged up to 25 years
Annual rate of change in eGFR (U25Crea) from the Week 8 to the Week 24 visit, including treatment effect extrapolation from (adult) EMPA-KIDNEY data | Up to week 24
Change from Day 1 to the Week 24 visit in urine protein-creatinine ratio (UPCR) | Up to week 24
The observed predose plasma concentrations of empagliflozin at the Week 26 visit | Up to week 26
Occurrence of at least one SAE or AE of special interest (AESI) per participant between Day 1 and the Week 24 visit, and between the Week 24 visit and end of treatment (EoT) +7 days residual effect period (REP) | Up to week 73
  SAE= serious adverse event AE= adverse event

CONTACTS AND LOCATIONS:
Locations (100):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford University Medical Center, Palo Alto, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Novak Center for Children's Health, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (3):
  - Hospital Italiano de Buenos Aires, CABA
  - Hospital de Niños Dr. Ricardo Gutierrez, CABA
  - Equipo Ciencia, CABA
- Australia (4):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Children's Hospital, Clayton, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
- Belgium (5):
  - HUB CHU Brugmann, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHC Mont Légia, Liège
- Canada (5):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
- France (6):
  - HOP Louis Pradel, Bron
  - HOP Timone, Marseille
  - HOP Enfants et Adolescents, Nantes
  - HOP Armand-Trousseau, Paris
  - Hôpital Necker, Paris
  - HOP des Enfants, Toulouse
- Germany (4):
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (3):
  - Semmelweis University, Faculty of Medicine, Budapest
  - University of Debrecen Clinical Centre, Debrecen
  - University of Pecs, Pécs
- Italy (4):
  - Istituto G. Gaslini, Genova
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Osp. Pediatrico Bambin Gesù, Roma
- Netherlands (5):
  - Amsterdam University Medical Center, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (5):
  - University Clinical Center, Gdansk, Gdansk
  - University Children's Hospital in Lublin, Lublin
  - L. Rydygier's Regional Hospital in Torun, Torun
  - The Children's Memorial Health Institute, Warsaw
  - University Clinical Hospital in Wrocław, Wroclaw
- Portugal (4):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULS de São José, E.P.E. - Hospital Dona Estefânia, Lisbon
  - ULS de Santa Maria, E.P.E, Lisbon
  - CHUP, EPE - Centro Materno Infantil do Norte, Porto
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Virgen del Rocío, Seville
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Karolinska University Hospital, Stockholm
- Turkey (Türkiye) (4):
  - Hacettepe University, Ankara
  - Ankara Universitesi Tip Fakultesi, Ankara
  - İstanbul Çapa University, Istanbul
  - Osmangazi University, Odunpazari
- United Kingdom (8):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - Great North Children's Hospital, Newcastle upon Tyne
  - Nottingham Children's Hospital, Nottingham
  - NIHR Southampton Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency